CLINICAL TRIAL: NCT01455753
Title: The Effect of Proximity on Flu-Shot Participation
Status: Completed | Type: Observational
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0006; P30AG034532 (NIH); P01AG005842 (NIH)
Record Dates: First submitted 2011-10-12; First posted 2011-10-20 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Influenza; Human
Keywords: Influenza; Proximity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Employees: A total of 1,801 employees of a health benefits administrator that held a free workplace influenza vaccination clinic.
  Interventions: Other: Functional Proximity; Other: Base Proximity

INTERVENTIONS:
Other: Functional Proximity — Using each employee's building entry/exit swipe card data, we test whether functional proximity-the likelihood that the employee walks by the clinic for reasons other than vaccination-predicts whether the employee gets vaccinated at the clinic.
Other: Base Proximity — We also test whether base proximity-the inverse of walking distance from the employee's desk to the clinic-predicts vaccination probability.

SUMMARY:
Using desk location information and employees' building entry/exit swipe card data from a company that offered a free 2-day worksite influenza vaccination clinic, we separately identify the vaccination effects of base proximity-the inverse of walking distance between one's desk and the clinic-and functional proximity-the likelihood of passing near the clinic during the course of a normal work day (ie, days when the clinic is not open).

DETAILED DESCRIPTION:
We study the 2011 influenza vaccine uptake of employees at the headquarters of a health benefits administrator in the United States. These employees are generally not health care personnel. All of them have health insurance. Of the company's total workforce (including those not based at the headquarters), 26% are African Americans and 37% are racial minorities.

There are 2 main buildings at the company headquarters. Building One houses 520 employees and is the site of the vaccination clinic; Building Two houses 1281 employees. The 2 buildings are 131 meters apart and connected by an enclosed passageway. The clinic was located near the cafeteria in Building One and adjacent to the passageway connecting the 2 buildings. The clinic was conducted from October 19 to 20, 2011, and it was advertised during the 3 weeks prior.

The company requires employees to swipe a personalized electronic badge to open the external doors of its buildings, which include the doors to the passageway between the buildings. The company provided us data on the date and time of each swipe in September and October 2011. If an employee swipes her badge and holds the door open for another employee, we do not observe that other employee. The badge swipe data are therefore an incomplete measure of all movements between the buildings. The company also gave us data on employee characteristics and vaccination uptake, scaled architectural plans of the buildings, and employee desk maps.

ELIGIBILITY:
Inclusion Criteria:

* Employee of Express Scripts.
* Eligible to receive a flu shot at Express Scripts.
* Over 18 years of age.

Exclusion Criteria:

* Children
* Non Express Scripts employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Employees at the headquarters of a health benefits administrator in the US. These employees are generally not health care personnel. All of them have health insurance.
  Of HQ employees, 520 are housed in Building 1 (the site of the vaccination clinic) and 1,281 are housed in Building 2. The two buildings are 131 meters apart and connected by an enclosed passageway. The clinic was located near the cafeteria in Building 1 and adjacent to the passageway connecting the two buildings.
Sampling Method: Non-Probability Sample
Enrollment: 1801 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Receipt of influenza vaccine | One week
  The investigators will measure whether proximity to a flu shot clinic effected whether an employee received an influenza vaccine.

SECONDARY OUTCOMES:
Absenteeism | The investigators will follow employees' absenteeism for five to six months
  The investigators will measure absenteeism in employees who received a flu shot versus employees who did not receive a flu shot.
Demographic characteristics on flu shot participation | Up to 3 years
  The investigators will explore how demographic characteristics correlate to employees receiving an influenza vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: David I Laibson, Ph.D., Principal Investigator — National Bureau of Economic Research, Harvard University
Locations (1):
- Express Scripts, St Louis, Missouri, United States

REFERENCES:
- [Result] Beshears J, Choi JJ, Laibson DI, Madrian BC, Reynolds GI. Vaccination Rates are Associated With Functional Proximity But Not Base Proximity of Vaccination Clinics. Med Care. 2016 Jun;54(6):578-83. doi: 10.1097/MLR.0000000000000523. PMID 27177295